CLINICAL TRIAL: NCT04485403
Title: The Effect of Ibuprofen on the Endocrine and Metabolic Status of Women With PCOS.
Brief Title: The Effect of Ibuprofen on Women With PCOS.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Beata Banaszewska, MD PhD Associate Proffesor Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 761/19
Record Dates: First submitted 2020-07-21; First posted 2020-07-24 (Actual); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: PCOS; Hyperandrogenism; Inflammation
Keywords: PCOS; IBUPROFEN; TESTOSTERON; HYPERANDROGENISM
MeSH Terms: conditions — Hyperandrogenism; Inflammation | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ibuprofen (Experimental): Depending on body weight, patients will be divided into two groups. Women with a body weight <70 kg will be taking a daily dose of 800 mg ibuprofen orally. Women ≥ 70 kg will take a dose of 1200 mg ibuprofen orally. Before and after 3 weeks of treatment, all subjects will have a full hormonal, biochemical and clinical profile.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — 800 mg/day ( 2 x 400mg) for 3 weeks in women with a bodyweight <70 kg, and a dose of 1200 mg/day (3x400mg) in women weighing> 70kg. The effects of treatment will be compared on the basis of changes in the hormonal profile and inflammatory markers, as well as the clinical assessment of the patient.

SUMMARY:
Polycystic ovary syndrome occurs in about 10% of women of childbearing age. His pathogenesis is not fully understood. More and more research concerns the role of chronic inflammation in these women as the cause of the disease. In vitro studies have shown a significant reduction in testosterone production by teak cells after ibuprofen. The goal of the project is to use a low dose of ibuprofen in women with PCOS to lower androgen levels.

DETAILED DESCRIPTION:
Polycystic ovary syndrome 1 is diagnosed in about 4-8% of women of childbearing age and is,therefore one of the most common endocrinopathies. The exact pathogenetic mechanism of PCOS is not fully discovered. Some women with PCOS have elevated levels of lutropin, which is considered to be the strongest stimulator of androgen production in ovarian theca cells. A breakthrough finding was the causal relationship between insulin resistance and hyperinsulinemia and hyperandrogenism in patients with PCOS. Confirmation of the theory that hyperinsulinemia is the cause of hyperandrogenism in these women gave the opportunity to treat women with PCOS by improving insulin sensitivity. The compartment of ovarian theca-interstitial cells is responsible for androgen overproduction in women with polycystic ovary syndrome. The cause of PCOS syndrome is seen in various mechanisms leading to the proliferation of thecal-interstitial cells. Factors that may affect the ovary in this way may include hyperinsulinemia, an increase in oxidative stress, exponents of generalized inflammation, and various cytokines such as TNF-alpha.

Prospective studies performed on women with polycystic ovary syndrome during perimenopause showed an increased incidence of type II diabetes, hypertension, ischemic heart disease, and myocardial infarction compared to the control group. In patients with PCOS, an abnormal, atherogenic lipid profile was found more often, characterized by increased total cholesterol, LDL and triglycerides, and decreased HDL fraction. Another risk factor for the development of cardiovascular disease are disorders in the functioning of vascular endothelial cells. In women with PCOS, elevated levels of C-reactive protein - a marker of chronic inflammation and endothelin-1, which are exponents of vascular endothelial disorders, were found. In addition, the risk of developing cardiovascular disease in women with PCOS is increased by elevated oxidative stress markers. Cardiometabolic diseases have been shown to be associated with abnormal vascular endothelial function and chronic inflammation. One of the most important and common indicators of inflammation is abnormally high levels of CRP. The acute phase protein is produced by hepatocytes due to stimulation by proinflammatory cytokines such as interleukin-6 (IL-6) and tumor necrosis factor (TNFα). Increased high sensitivity CRP (hs-CRP) is considered to be one of the most important predictors of the risk of cardiovascular events. In addition to C-reactive protein, inflammatory cytokines and chemokines, including IL-18, monocyte-1 chemotactic protein (MCP-1) and macrophage-1a inflammatory protein (MIP-1a) play an important role in chronic inflammation. Interleukin-18 appears to be associated with insulin resistance and metabolic syndrome and has prognostic value for cardiovascular death. An increased C-reactive protein concentration was found in the group of women with PCOS. In 2011, the latest meta-analysis confirming the increased concentration of hsCRP was presented. Increased IL-18 levels were observed in women with polycystic ovary syndrome, which correlated with obesity and total testosterone levels. Individual studies have also shown an increase in the concentration of monocyte-1 chemotactic protein (MCP-1) in these women. In 2005, Orio et al. Showed a significantly elevated white blood cell (WBC) concentration in a group of 150 women with PCOS. Oxidative stress and chronic inflammation are closely related and form a vicious circle concept in which inflammation generates reactive oxygen species (ROS), while oxidative stress promotes and exacerbates inflammation. The first report documenting increased oxidative stress in women with PCOS was published in 2001 by Sabuncu. It was assessed by lipid peroxidation, which was significantly higher in PCOS and positively correlated with BMI, insulin concentration and blood pressure. In reference to these risks for women with PCOS - last, the latest and most arousing emotions pathogenetic theory this team is chronic inflammation probably caused by the improper composition of bacterial microflora microbiota. However, there are many undiscovered interrelationship mechanisms between inflammation and endocrine disorders. One of the theories may be the role of lipopolysaccharide (LPS) released from Gram (-) bacteria and adversely affecting metabolic functions, and above all insulin resistance. In 2012, a paper was published in which a correlation between LPS binding protein and metabolic syndrome and inflammatory markers was demonstrated. The second hypothesis is the induction of chronic inflammation through specific pathogens. Microorganisms such as Chlamydia pneumoniae and Helicobacter pylori are associated with chronic inflammation and cardiovascular disease. In particular, Chlamydia pneumoniae infection correlates with the presence of atherosclerosis and even acute myocardial infarction, and chronic inflammatory processes associated with periodontal disease are associated with cardiovascular risk. The theory of specific microorganisms probably remains the most controversial and least studied concept between PCOS and chronic infection. Morin-Papunen et al. Observed a higher amount of IgG Chlamydia pneumonia and Chlamydia trachomatis and hsCRP in women with no ovulation and hirsutism than in the control group. In another study, the amount of Helico-bacterial pylori was more common in women with PCOS than in the age-matched control group. In 2011, Dursun published a paper on periodontal infection in women with PCOS compared to a control group of the same age and comparable body weight.

The new hypothesis for the treatment of polycystic ovarian syndrome is based on the assumption that ibuprofen inhibits the proliferation of ovarian theca-intestinal cells, lowers streroidogenesis, and additionally has a positive effect on insulin and reduces oxidative stress. Ibuprofen is a medicament from the group of NSAID used for the purpose of reducing the state zap a cast and analgesic dosage depends on the indication and the patient's condition. For non-prescription oral ibuprofen, the maximum daily dose is 1.2 g and has a good safety profile. Under the supervision of a physician and on his behalf, in some indications, higher doses are used, even up to 3.2 g per day. Low risk of gastrointestinal, hepatorenal and other complications has been demonstrated. Some, but not all, studies show a slightly increased cardiovascular risk, but in general, all complications occur less frequently than when using diclofenac or coxib. Ibuprofen in over-the-counter doses has a low risk of serious gastrointestinal (GI) complications and the development of kidney problems and heart disease. Irreversible liver damage is not observed in patients using it, as it sometimes occurs in patients using paracetamol or aspirin.

The use of ibuprofen in women with PCOS may improve the endocrine and metabolic profile which may reduce the risk associated with cardiovascular disease

The mechanisms of action of ibuprofen that gave rise to use in the treatment of PCOS are as follows :

In vitro Ibuprofen inhibits the genes that regulate androgen production ( CYP11 , CYP17 and HSD ) Ibuprofen inhibits the expression of key genes regulating androgen synthesis by IL-1β and LPS Ibuprofen attenuates the stimulating effect of IL-1β on the growth of theca cells

Project goals A. Assessment of the effect of ibuprofen on the endocrine and metabolic profile in women with PCOS B. The effect of ibuprofen on chronic inflammation in women with PCOS

C Recruitment of the patients for testing is scheduled for a period of one year. Will be based on the classification of patients into three-week application of the ibuprofen, and assessing the effects of the use of this drug in the daw which 8 00 mg/day ( 2 x 4 00mg) for 3 weeks in women with a bodyweight <70 kg, and a dose of 1200 mg/day (3x400mg) in women weighing> 70kg. The effects of treatment will be compared on the basis of changes in the hormonal profile and inflammatory markers, as well as the clinical assessment of the patient.

ELIGIBILITY:
Inclusion Criteria (patient should meet all the criteria)

1. Diagnosis of PCOS according to Rotterdam Criteria
2. Written consent to participate in a clinical trial
3. Age up to 40 years
4. Irregular periods (> 35 days) or secondary amenorrhea over 3 months
5. Hyperandrogenism (hirsutism and / or acne) and / or total serum testosterone> 0.5 ng / mL

Exclusion Criteria:

1. A diagnosed chronic disease, including in particular:

   * Cancer of the ovary, adrenal gland, endometrium, cervix, mammary gland
   * Congenital adrenal hyperplasia (17-OH- progesterone> 2 ng / mL)
   * Clinically diagnosed Cushing's disease, acromegaly, gigantism
   * Type I or II diabetes
   * Gastrointestinal diseases (peptic ulcer, inflammatory bowel disease, liver disease)
   * Active or history of gastric and duodenal ulceration, perforation or bleeding, also following NSAIDs. Gastrointestinal bleeding
   * Severe hepatic impairment, severe renal insufficiency or severe heart failure.
   * Hemorrhagic diathesis.
   * systemic lupus erythematosus and mixed connective tissue disease
   * a history of hypertension and cardiac dysfunction
   * kidney problems
2. Unexplained vaginal bleeding
3. Use of hormonal treatment currently or during the last 2 months
4. Unexplained abdominal pain
5. Chronic use of drugs, especially: lithium salts, warfarin, oral hypoglycaemics, contraceptives, methotrexate, drugs that lower blood pressure, ACE inhibitors, b-blockers, diuretics that may cause interactions with ibuprofen, corticosteroids, mifepristone,
6. Hypersensitivity to ibuprofen or any of the excipients.
7. Existing or past allergy symptoms in the form of a runny nose, urticaria or bronchial asthma after taking acetylsalicylic acid or other non-steroidal anti-inflammatory drugs., Cyclosporin, quinoline antibiotics
8. Pregnancy and lactation
9. Concomitant use of other nonsteroidal anti-inflammatory drugs, including selective COX-2 inhibitors (increased risk of side effects).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Decrease of Testosteron levels | 3 weeks
  total testosterone level measurement

SECONDARY OUTCOMES:
Decrease in hyperandrogenism markers | 3 weeks
  hirsutism evaluation ( Ferriman-Gallway score, acne evaluation, androstendion, DHEA-S, SHBG level evaluation)

OTHER OUTCOMES:
Influence of ibuprofen on the decrease chronic inflammatory state in PCOS patients | 3 weeks
  hsCRP

CONTACTS AND LOCATIONS:
Overall Officials: Beata Banaszewska, Principal Investigator — Poznan University of Medical Sciences, Poland
Locations (1):
- Division of Infertility and Reproductive Endocrinology, Department of Gynecology and Obsterics, Poznan, Greater Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No